CLINICAL TRIAL: NCT06073418
Title: Dietary Habits, Nutritional Knowledge and Physical Activity Assessment in Early Stage Breast Cancer Patients (DEMETRA)
Brief Title: Dietary Habits, Nutritional Knowledge and Physical Activity Assessment in Early Stage Breast Cancer Patients
Acronym: DEMETRA
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2022-30
Record Dates: First submitted 2023-09-01; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The advances in early detection coupled with improvements in treatments have led to an ever increasing number of breast cancer survivors. New methods to improve outcomes, including strategies aimed at improving the quality of life and reducing the risk of other diseases, may complement the currently available treatment options. In particular, interventions targeting diet, weight and physical activity can reduce the risk of cancer occurrence, prevent cancer recurrence, and improve survival and the quality of life.This cross-sectional, prospective, observational study aims at evaluating dietary habits and nutritional knowledge in patients with early hormone receptor positive and hormone receptor negative breast cancer.

DETAILED DESCRIPTION:
The advances in early detection coupled with improvements in treatments have led to an ever increasing number of breast cancer survivors. New methods to improve outcomes, including strategies aimed at improving the quality of life and reducing the risk of other diseases, may complement the currently available treatment options. In particular, interventions targeting diet, weight and physical activity can reduce the risk of cancer occurrence, prevent cancer recurrence, and improve survival and the quality of life.

The Women's Intervention Nutrition Study (WINS) and the Women's Healthy Eating and Living (WHEL) Randomized Trial examined the impact of dietary intervention on disease outcome in patients with early stage breast cancer, but with different results.

The Women's Intervention Nutrition Study randomized 2437 women with early stage breast cancer to receive a low-fat dietary intervention or usual care control and it demonstrated that dietary intervention improves disease free-survival of breast cancer patients receiving conventional cancer management. Although these benefit was no longer statistically significant at a longer follow-up, an exploratory subgroup analysis revealed that patients with hormone receptor-negative breast cancer continued to experience benefits from the intervention.

The Women's Healthy Eating and Living (WHEL) Randomized Trial, randomized 3088 women previously treated for early breast cancer, to receive low-fat, high-fruit, vegetable and fiber diet or to the control group. This trial failed to demonstrate a benefit in terms of recurrence rates within the experimental group.

Given the discrepancies among the findings of these two large trials, dietary changes are not routinely suggested as part of adjuvant therapies for breast cancer survivors and further research is needed to expand knowledge in this area. This study aims at evaluating dietary habits and nutritional knowledge in patients with early hormone receptor positive and hormone receptor negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgically removed early stage (I-IIIa) hormone receptor-positive or hormone receptor negative breast cancer. Patients with hormone receptor-positive breast cancer can be in treatment with endocrine therapy; patients with hormone receptor-negative tumors have to be in follow-up. Concomitant use of targeted therapies with anti-hormonal agents is allowed only in adjuvant setting
* Female patients ≥18 years of age.
* Written informed consent must be obtained before any study-related assessment is performed

Exclusion Criteria:

* Patients with advanced/metastatic breast cancer.
* Patients with early breast cancer receiving (neo)adjuvant chemotherapy or anti-HER2 agents
* Patients receiving active treatment for secondary primary tumors (excluding basal cell carcinoma or in situ neoplasias)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with early stage hormone receptor positive breast cancer treated at the Department of Medical Oncology and Cancer Prevention, IRCCS National Cancer Institute of Aviano and at the other involved clinical centers considered eligible for the study will be enrolled, after providing written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 1098 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2032-07-01 (Estimated); Study Completion 2032-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of nutritional knowledge in patients with surgically removed early breast cancer | At baseline and at 3-5 years of follow up
  Median and interquartile range of items of nutritional knowledge questionnaire in patients with surgically removed early breast cancer
Evaluation of dietary habits in patients with surgically removed early breast cancer | At baseline and at 3-5 years of follow up
  Frequency of different answers at dietary habits questionnaire
Evaluation of physical activity in patients with surgically removed early breast cancer | At baseline and at 3-5 years of follow up
  Frequency of different answers at activity questionnaire

SECONDARY OUTCOMES:
Association between nutritional knowledge and physical activity | At baseline and at 3-5 years of follow up
  difference in nutritional knowledge score between subgroups of patients with different levels of physical activity
Association between nutritional knowledge and dietary habits | At baseline and at 3-5 years of follow up
  difference in nutritional knowledge score between subgroups of patients with different frequencies of consumption for selected foods
Association between dietary habits and physical activity | At baseline and at 3-5 years of follow up
  association between frequencies of consumption for selected foods and levels of physical activity
Association between dietary habits and BMI | At baseline and at 3-5 years of follow up
  Difference in frequencies of consumption for selected foods between BMI categories
Association between dietary habits and waist to hip ratio | At baseline and at 3-5 years of follow up
  Difference in mean of waist to hip ratio between subgroups of patients with different frequencies of consumption for selected foods
Association between dietary habits and anthropometric measure | At baseline and at 3-5 years of follow up
  Difference in mean of waist, hip, abdomen circumferences between subgroups of patients with different frequencies of consumption for selected foods
Association between dietary habits and blood tests results | At baseline and at 3-5 years of follow up
  Differences in mean level of selected blood test (e.i glycemia, HDL, LDL) between subgroups of patients with different frequencies of consumption for selected foods
Association between dietary habits and disease relapse | From baseline up to 5 years of follow up
  Association between answers to dietary habits questionnaire and progression free survival defined as the time from study enrolment until progression or death from any cause whichever comes first
Association between dietary habits and overall survival | From baseline up to 5 years of follow up
  Association between answers to dietary habits questionnaire and overall survival defined as the time from study enrolment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Mattia Garutti, MD, Principal Investigator — IRCCS-Centro di Riferimento Oncologico (CRO), Aviano (PN)
Locations (1):
- IRCCS, Centro di Riferimento Oncologico (CRO) di Aviano, Aviano, Pordonone, Italy